CLINICAL TRIAL: NCT04834011
Title: Complete Mesocolic Excision (CME) and Central Vascular Ligation (CVL) in Right-sided Colon Cancer: Surgical and Radiological Assessment. A Prospective Observational Study (RACOMERC)
Brief Title: Radiologic Assessment in Complete Mesocolic Excision for Right Colon Cancer (RACOMERC)
Acronym: RACOMERC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof. Antonino Agrusa, Associate professor, University of Palermo
Other Study IDs: RACOMERC 01/2021
Record Dates: First submitted 2021-03-22; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Right-sided Colon Cancer
Keywords: Right colon cancer; complete mesocolic excision; CT abdominal scan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Laparoscopic right colonic resection with Complete Mesocolic Excision (CME)
Radiation: 3D CT angiography

SUMMARY:
Colorectal surgery has made progressive advances in recent years related on one hand to the implementation of diagnostic methods that allow an early diagnosis of tumors and on the other hand to the development of therapeutic options based on laparoscopic surgery. In particular, multicenter clinical trials have shown that the laparoscopic approach to colorectal cancer had a comparable or even better outcomes in terms of perioperative complications and functional recovery of patients than traditional surgery. Complete Mesocolic Excision (CME) in right colonic resections is a surgical approach, of greater technical complexity, that appears to improve the oncological outcomes of these patients at the cost of an increased rate of complications. The highest rate of complications reported in the literature in patients undergoing CME was related to intraoperative bleeding due to the central vascular dissection that is performed. CT technological advances have made possible to perform CT angiography with multiplanar and three-dimensional reconstructions with the possibility of obtaining a detailed preoperative map of the vascular anatomy of these patients. CT scan was acquired immediately before contrast material injection and during arterial and venous phase. Arterial phase was obtained using the bolus tracking technique with an automated scan-triggering software. Image analysis was performed using multiplanar reformations (MPR), maximum intensity projection (MIP) and 3D volume rendering (VR) technique. The purpose of the CT was to identify three different parameters necessary for proper performance of CME and CVL and to compare preoperative observations with intraoperative evidence. All surgeries were performed by teams experienced in laparoscopic colorectal surgery. The investigators evaluated:- Fascia of Fredet; vascular structures; lymph nodes.

DETAILED DESCRIPTION:
x

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of right-sided colon cancer
* patients underwent to CT angiography
* laparoscopic right hemicolectomy with CME and CVL.

Exclusion Criteria:

* metastatic disease
* palliative treatment
* impossibility to perform CT angiography
* patients underwent to a traditional colonic resection with D2 lymphadenectomy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with endoscopic diagnosis of right-sided colon cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Preoperative radiologic assessment of patients with diagnosis of right-sided colon cancer. The investigators evaluated: fascia of Fredet; vascular structures (ileocolic vessels; right colic artery, middle colic artery, trunk of Henle); lymph nodes. | Evaluation of preoperative CT scan features during enrollment of patients.
  Evaluation of preoperative CT scan features during enrollment of patients.

SECONDARY OUTCOMES:
Perioperative outcomes: intraoperative complications | intraoperative time
  complication occurred during surgery
Perioperative outcomes: postoperative complications | up to 30 days postoperative
  complication occurred in postoperative period
Perioperative outcomes: mean operative time | intraoperative time
  operative time
perioperative outcomes: rate of conversion | intraoperative time
  rate of conversion from laparoscopy to open surgery

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Agrusa, Professor, Principal Investigator — University of Palermo - Italy
Locations (1):
- Azienda Ospedaliera Universitaria Policlinico "P. Giaccone" Palermo - University of Palermo, Palermo, Italy - Sicily, Italy

REFERENCES:
- [Background] Mike M, Kano N. Laparoscopic surgery for colon cancer: a review of the fascial composition of the abdominal cavity. Surg Today. 2015 Feb;45(2):129-39. doi: 10.1007/s00595-014-0857-9. Epub 2014 Feb 11. PMID 24515451
- [Background] Mari FS, Nigri G, Pancaldi A, De Cecco CN, Gasparrini M, Dall'Oglio A, Pindozzi F, Laghi A, Brescia A. Role of CT angiography with three-dimensional reconstruction of mesenteric vessels in laparoscopic colorectal resections: a randomized controlled trial. Surg Endosc. 2013 Jun;27(6):2058-67. doi: 10.1007/s00464-012-2710-9. Epub 2013 Jan 5. PMID 23292563
- [Background] Acar HI, Comert A, Avsar A, Celik S, Kuzu MA. Dynamic article: surgical anatomical planes for complete mesocolic excision and applied vascular anatomy of the right colon. Dis Colon Rectum. 2014 Oct;57(10):1169-75. doi: 10.1097/DCR.0000000000000128. PMID 25203372
- [Background] Murono K, Kawai K, Ishihara S, Otani K, Yasuda K, Nishikawa T, Tanaka T, Kiyomatsu T, Hata K, Nozawa H, Yamaguchi H, Watanabe T. Evaluation of the vascular anatomy of the right-sided colon using three-dimensional computed tomography angiography: a single-center study of 536 patients and a review of the literature. Int J Colorectal Dis. 2016 Sep;31(9):1633-8. doi: 10.1007/s00384-016-2627-1. Epub 2016 Jul 27. PMID 27461539
- [Background] Miyazawa M, Kawai M, Hirono S, Okada K, Shimizu A, Kitahata Y, Yamaue H. Preoperative evaluation of the confluent drainage veins to the gastrocolic trunk of Henle: understanding the surgical vascular anatomy during pancreaticoduodenectomy. J Hepatobiliary Pancreat Sci. 2015 May;22(5):386-91. doi: 10.1002/jhbp.205. Epub 2015 Jan 7. PMID 25565654